CLINICAL TRIAL: NCT03581305
Title: PET Imaging of the Dopaminergic and Serotonergic Systems in Treated HIV Positive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 180117; 18-CC-0117 (Other: NIH protocol number)
Record Dates: First submitted 2018-07-07; First posted 2018-07-10 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-04-07

CONDITIONS: Depression; HIV Infections; HIV-Associated Cognitive Motor Complex
Keywords: 11C-DASB; 18F-Fluoro-L-dopa; HIV; Depression; Positron Emission Tomography (PET)
MeSH Terms: conditions — Depression; HIV Infections; AIDS Dementia Complex | interventions — fluorodopa F 18; 3-amino-4-(2-dimethylaminomethylphenylsulfanyl)benzonitrile

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dopaminergic arm (Active Comparator): 25 eligible HIV-infected individuals and 50 eligible HIV-negative (HIV-) individuals for the dopaminergic arm.
  Dopaminergic arm:
  Group A: HIV-positive subjects with or without co- morbidities; Group B: HIV-negative subjects with co-morbidities; Group C: HIV-negative subjects without co-morbidities
  Interventions: Drug: 18F-FDOPA
- Serotonergic arm (Active Comparator): 20 HIV-infected individuals and 20 HIV-negative individuals for the serotonergic arm
  Serotonergic arm:
  Group D: HIV-positive subjects with or without co-morbidities; Group E: HIV-negative subjects with or without co-morbidities
  Interventions: Drug: 11C-DASB

INTERVENTIONS:
Drug: 18F-FDOPA — High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
  Arms: Dopaminergic arm
Drug: 11C-DASB — High resolution positron emission tomography (PET) of the brain and radioligands targeted against the serotonergic (11C-DASB) system.
  Arms: Serotonergic arm

SUMMARY:
Background:

Human immunodeficiency virus (HIV) infection is a serious disease with no cure. Some people with HIV have depression and other mood problems. They can have problems with thinking and memory. Researchers think 2 chemicals in the brain may cause those problems. The chemicals are serotonin and dopamine. The researchers want to take images to learn more about those chemicals in HIV patients.

Objective:

To learn how HIV affects serotonin and dopamine in the brain.

Eligibility:

Adults ages 18-70 with HIV who have been on antiretroviral treatment for at least 1 year

Healthy adults ages 18-70

All participants must be already enrolled in protocol 13-N-0149.

Design:

* Participants will be screened with a urine drug test. The results could be shared with insurance companies.
* Participants who could be pregnant will have a pregnancy test.
* Participants may have a physical exam and blood tests.
* Participants will have 1 or 2 positron emission tomography (PET) scans. A needle will guide a thin plastic tube (catheter) into an arm vein. A radioactive drug will be injected into the plastic tube. This is a tracer that helps researchers understand the PET images.
* Participants who have the dopamine scan will have to fast for 4-6 hours before the scan. They will take a pill to help direct the tracer to the brain one hour before the scan.
* Each scan will last about 1.5 hours.
* Participants will be asked to drink a lot of fluids and empty their bladder frequently for the rest of the day after each scan.

DETAILED DESCRIPTION:
Background: An extensive body of literature points towards neuronal brain injury in human immunodeficiency virus positive (HIV-positive) subjects despite virological suppression of the virus in the periphery under the effect of antiretroviral therapies (ART). Existing evidence suggests that the central nervous system (CNS) could be an important reservoir for human immunodeficiency virus (HIV) regardless of cumulative time on treatment. This results in progressive neurocognitive dysfunction despite optimal treatment and peripheral control of the infection. Even though structural imaging studies have described abnormalities in optimally-treated HIV-positive subject population, there has been only a few attempts at deciphering the cellular levels of brain damage in those subjects using in vivo molecular imaging biomarkers. As part of CNS involvement, specific neurotransmitter systems including the dopaminergic and serotonergic systems are thought to be affected by the infection with distinct neurological, cognitive and psychological manifestations, even in optimally-treated subjects.

Objective: This protocol aims at identifying aspects of dopaminergic and serotonergic dysfunction in optimally-treated HIV-positive subjects using high resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) and serotonergic (11C-DASB) systems.

Study population: We will identify 25 eligible HIV-infected individuals and 50 eligible HIV-negative (HIV-) individuals for the dopaminergic arm, and 20 HIV-infected individuals and 20 HIV-negative individuals for the serotonergic arm. Subjects will be selected from IRB approved NIH protocols, self-referred or will be referred form outside providers/institutions and those who meet eligibility criteria will be offered enrollment in our study.

Design: Subjects will undergo either a one-time 18F-FDOPA PET scan or a one-time 11C-DASB PET scan or both, if eligible. HIV-positive subjects and HIV-negative individuals will be included in the study.

Outcome Measures: Influx constant (Ki) for 18F-FDOPA PET and Binding potential relative to

non-displaceable binding (BPND) values for 11C-DASB PET

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject groups:

* Dopaminergic arm:

  * Group A: HIV-positive subjects with or without co-morbidities
  * Group B: HIV-negative subjects with co-morbidities
  * Group C: HIV-negative subjects without co-morbidities
* Serotonergic arm:

  * Group D: HIV-positive subjects with or without co-morbidities
  * Group E: HIV-negative subjects with or without co-morbidities

All Subjects (Groups A-E):

1. Men and women, 18-70 years of age
2. Ability to sign informed consent by the subject
3. Subjects may be enrolled in or have been discharged from IRB approved NIH protocols OR subjects may be referred from outside providers/institutions.
4. Has the ability to be seen by an outside medical doctor who provides care.

All HIV-positive Subjects with or without co- morbidities (Groups A [dopaminergic arm, n=25)] and Group D [serotonergic arm, n=20])

1. Known and documented HIV-1 infection
2. Plasma HIV-RNA BLD (<100 copies/mm3) for greater than one year since the last available documented viral load measurement..
3. At least one year of continuous ART prior to last documented suppressed viral load measurement and no history of ART modification or interruption since then.

HIV-negative Subjects WITH Co-morbidities (Group B, n=25)

1. HIV-antibody negative
2. At least one or more of the following criteria:

   1. Hypertension, as defined by treatment with medications for hypertension or with a systolic blood pressure at screening greater than or equal to 140mm Hg.
   2. Diabetes mellitus, as defined by HgbA1C greater than or equal to 6.5% or known treatment for diabetes.
   3. Hepatitis C infection as documented by lab results of a positive Hepatitis C antibody and/or detectable Hepatitis C viral load. Subjects who responded to HCV treatment (SVR) will be included.
   4. History of previous but not current drug abuse.
   5. History of previous but not current alcoholism (defined as alcohol intake that affect/affected the subject s work or home life).
   6. Clinical atherosclerotic cardiovascular disease (ASCVD) (e.g. history of acute coronary syndromes, or myocardial infarction, stable or unstable angina, coronary or other arterial revascularization or peripheral arterial disease of atherosclerotic origin) and/or 10-year heart disease risk score (ASCVD risk score) >7.5% (7.5 % score is the threshold for starting statin therapy as per the 2013 American College of Cardiology [ACC] / American Heart Association [AHA] guidelines).

HIV-negative Subjects WITHOUT co-morbidities (Group C, n=25)

1. HIV-antibody negative
2. No history of any of the following:

   1. Hypertension, as defined by treatment with medications for hypertension or with a systolic blood pressure at screening greater than or equal to 140mm Hg.
   2. Diabetes mellitus, as defined HgbA1C greater than or equal to 6.5% or treatment for diabetes.
   3. Hepatitis C infection as documented by lab results of positive Hepatitis C antibody and/or detectable Hepatitis C viral load. Subjects who responded to HCV treatment (SVR) will not be included.
   4. History of previous drug abuse.
   5. History of previous alcoholism. Alcoholism is based on alcohol having affected the subject s work or home life.
   6. Clinical ASCVD (e.g. history of acute coronary syndromes, or myocardial infarction, stable or unstable angina, coronary or other arterial revascularization or peripheral arterial disease of atherosclerotic origin) and/or 10-year heart disease risk score (ASCVD risk score) >7.5% (7.5 % score is the threshold for starting statin therapy as per the 2013 ACC/AHA guidelines 35).
   7. Any other disease entities including chronic infections (e.g. Hepatitis B, Lyme disease), neurological diseases (e.g. Multiple sclerosis, vasculitis) or systemic diseases (e.g. Sjogren s diseases, sarcoidosis, systemic lupus erythematosus [SLE]) that in the opinion of the investigator would be considered a significant co-morbidity.

HIV-negative Subjects with or without co- morbidities (Group E, n=20)

1. HIV-antibody negative

EXCLUSION CRITERIA:

All Subjects (Groups A-E):

1. Illness or other condition that, in the opinion of the PI, may interfere with study participation at the time of enrollment, including known history of significant intracranial structural damage such as previous stroke(s) or history of intracranial benign or malignant tumors.
2. Conditions other than HAND associated with cognitive impairment or dementia such as Alzheimer s, Parkinson s disease, head injury with loss of consciousness >30 minutes, or seizure disorders.
3. A positive screening result for psychiatric diseases that are known to affect the dopaminergic or serotonergic systems.
4. Current substance abuse that would interfere with PET scan results at the investigators discretion.
5. Medications: use of any drug with known dopaminergic or serotonergic activity within 6 months prior to planned imaging date(s).
6. Pregnant or Lactating women: Women of childbearing potential must have a negative serum or urine pregnancy test within 1 week prior to study entry. Pregnancy testing will also be performed in enrolled female participants prior to any radiation exposure.
7. Prior or planned/anticipated exposure to radiation due to clinical care or participation in other research protocols, which would exceed the recommended acceptable annual limit of radiation exposure once accounting for the requirements of the current study.

Additional Exclusion Criteria for the Dopaminergic Arm (Groups A, B and C):

1. Use of any of the following drugs within 6 months from planned imaging date(s):

   1. Haloperidol (increased intracerebral dopamine turnover caused by haloperidol may result in increased accumulation of 18F-DOPA)
   2. Monoamine oxidase (MAO) inhibitors (may result in increased accumulation of 18F-DOPA in the brain)
   3. Reserpine (reserpine-induced depletion of the contents of intraneuronal vesicles may prevent retention of 18F-DOPA in the brain)
   4. Carbidopa/LDOPA (LDOPA competes with 18F-DOPA for DOPA decarboxylase activity)
2. Allergy to carbidopa

Note that HBV is not an exclusion criterion for groups A, B, D or E since it s not known to have direct CNS pathology in the absence of advanced liver disease and cirrhosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dima A Hammoud, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
No plan for sharing IPD

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-CC-0117.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through protocol number 13-N-0149, other IRB- approved intramural NIH protocols, or through referrals from outside providers/ institutions or self-referred. Once consented and found eligible, subjects underwent PET scanning using 18FDOPA and / or 11C-DASB. All visits were on a outpatient basis. There were not follow-up visits after the completion of the PET scan(s) The recruitment and enrollment process for this study occurred from 11/20/2018 through 11/5/2021
Pre-assignment Details: Among HIV positive subjects:
  1 subject didn't show up to either scan 2 subjects couldn't finish FDOPA and didn't come back for DASB 2 subjects did FDOPA but didn't come back for DASB
  Among HIV negative subjects
  1 subject did DASB but didn't come back for FDOPA
Groups:
- HIV Positive Participants: * 25 eligible HIV-infected participants for the dopaminergic arm Plan: 18F-FDOPA PET: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
  * 20 HIV-infected individuals for the serotonergic arm Plan: 11C-DASB: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the serotonergic (11C-DASB) system.
- HIV Negative Participants: * 50 eligible HIV-negative participants for the dopaminergic arm Plan: 18F-FDOPA PET: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
  * 20 HIV-negative participants for the serotonergic arm Plan: 11C-DASB: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the serotonergic (11C-DASB) system.
Period: Dopaminergic Study
Arm/Group | HIV Positive Participants | HIV Negative Participants
Started | 23 | 23
Completed (this includes participants who finished the scan) | 20 | 22
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — could not finish FDOPA scan | 2 | 0
Period: Serotonergic Study
Arm/Group | HIV Positive Participants | HIV Negative Participants
Started (this includes participants who finished the DASB scan.) | 23 | 23
Completed | 18 | 22
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Population: All participants in the dopaminergic and serotonergic arms, irrespective of study completion, based on HIV status
Groups:
- HIV Positive Participants (Dopaminergic and Serotonergic Studies): 25 eligible HIV-infected individuals for the dopaminergic arm
  18F-FDOPA: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
  20 eligible HIV-infected individuals for the serotonergic arm
  11C-DASB: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the serotonergic (11C-DASB) system.
- HIV Negative Participants (Dopaminergic and Serotonergic Studies): 50 eligible HIV-negative (HIV-) individuals for the dopaminergic arm
  18F-FDOPA: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
  20 eligible HIV-negative individuals for the serotonergic arm
  11C-DASB: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the serotonergic (11C-DASB) system.
- Total: Total of all reporting groups
Arm/Group | HIV Positive Participants (Dopaminergic and Serotonergic Studies) | HIV Negative Participants (Dopaminergic and Serotonergic Studies) | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants] — Population: those are the screened participants who completed the study (participants in either the serotonergic or dopaminergic studies or both) separated by HIV status
  Participants
    number analyzed (Participants) | 20 | 23 | 43
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 18 | 21 | 39
    >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Those are the participants who completed the study (either the serotonergic or dopaminergic studies or both) separated by HIV status
  Participants
    number analyzed (Participants) | 20 | 23 | 43
    Female | 6 | 9 | 15
    Male | 14 | 14 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Those are the participants who completed the study (either the serotonergic or dopaminergic studies or both) separated by HIV status
  Participants
    number analyzed (Participants) | 20 | 23 | 43
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 9 | 13 | 22
    White | 11 | 10 | 21
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
participant numbers [Count of Participants; unit: Participants] — Population: Those are the participants who completed either the serotonergic or dopaminergic studies or both, separated by HIV status
  Participants
    number analyzed (Participants) | 20 | 23 | 43
    (all) | 20 | 23 | 43

OUTCOME MEASURES:

1. Primary Outcome: Influx Constant (Ki) for 18F-FDOPA PET.
Description: in order to learn how HIV affects dopamine in the brain, we performed dynamic PET scans for 90 minutes in each patient, after injection of FDOPA.
  Analysis: After the scans were reconstructed, we extracted the Time activity curves and performed compartmental analysis using Patlak linear graphical analysis with reference region.
  The extracted outcome measure is the influx constant referred to as Ki and reflecting the rate of FDOPA uptake in specific brain regions.
Time Frame: 90 minutes of scanning
Population: All participants who completed FDOPA PET scan with usable Data
Measure: Mean (Standard Deviation); unit: min-1
Groups:
- Dopaminergic Arm Group A: 25 eligible HIV-infected individuals for the dopaminergic arm.
  Dopaminergic arm:
  Group A: HIV-positive subjects with or without co- morbidities;
  18F-FDOPA: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
- Dopaminergic Arm Group B/C: 50 eligible HIV-negative (HIV-) individuals for the dopaminergic arm.
  Group B: HIV-negative subjects with co-morbidities; Group C: HIV-negative subjects without co-morbidities
  18F-FDOPA: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
Arm/Group | Dopaminergic Arm Group A | Dopaminergic Arm Group B/C
Number analyzed (Participants) | 19 | 20
min-1
  Caudate | 0.01415 (0.00136) | 0.01409 (0.00126)
  Putamen | 0.01588 (0.00127) | 0.01592 (0.00127)

2. Primary Outcome: 11C-DASB PET Binding Potential
Description: Binding potential is a measure of the density of available serotonin transporter in specific brain locations. This is extracted from time activity curves of dynamic PET data acquired over 90 minutes after injection of 11C-DASB.
Time Frame: 90 minutes of scanning
Measure: Mean (Standard Deviation); unit: unitless
Groups:
- Serotonergic Arm Group D: IRB approved numbers:
  20 eligible HIV-infected individuals
  final analyzed numbers:17 participants with good quality PET scans and within normal limits neuropsychological testing
- Serotonergic Arm Group E: IRB approved numbers:
  20 eligible HIV-negative (HIV-) individuals
  final analyzed number: 19 participants with good quality PET scans and within normal limits neuropsychological testing
Arm/Group | Serotonergic Arm Group D | Serotonergic Arm Group E
Number analyzed (Participants) | 17 | 19
unitless | 2.949 (0.395) | 3.256 (0.597)

3. Secondary Outcome: Correlation of 18F-FDOPA With Co-morbidities
Description: Correlation of 18F-FDOPA uptake in the brain with co-morbidities such as cardiovascular disease
Time Frame: Study and statistical analysis Completion
Reporting Status: Not Posted, anticipated posting 2023-06

4. Secondary Outcome: Correlation of 18F-FDOPA and 11C-DASB With HIV
Description: Correlation of 18F-FDOPA and 11C-DASB with HIV infection parameters (e.g. time since HIV diagnosis, duration of infection before treatment initiation, nadir CD4).
Time Frame: Study and statistical analysis Completion
Reporting Status: Not Posted, anticipated posting 2023-06

5. Secondary Outcome: Correlation of 11C-DASB With Neuropsychiatric Evaluation
Description: Correlation of 11C-DASB with Neuropsychiatric evaluation (e.g. depressive and executive function/cognitive scores).
Time Frame: Study and statistical analysis Completion
Reporting Status: Not Posted, anticipated posting 2023-06

ADVERSE EVENTS:
Time Frame: 90 minutes of scanning
Description: the definition of adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the clinicaltrials.gov
Groups:
- HIV Positive Subjects: 25 eligible HIV-infected individuals for the dopaminergic arm
  18F-FDOPA: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
  20 HIV-infected individuals for the serotonergic arm
  11C-DASB: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the serotonergic (11C-DASB) system.
- HIV Negative Subjects: 50 eligible HIV-negative individuals for the dopaminergic arm
  18F-FDOPA: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the dopaminergic (18F-FDOPA) system.
  20 HIV-infected individuals and 20 HIV-negative individuals for the serotonergic arm
  11C-DASB: High resolution positron emission tomography (PET) of the brain and radioligands targeted against the serotonergic (11C-DASB) system.
Arm/Group | HIV Positive Subjects | HIV Negative Subjects
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT03581305/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03581305/ICF_001.pdf